CLINICAL TRIAL: NCT04210453
Title: The Impact of Vitamin C on Postoperative Acute Kidney Injury in Risk Patients Undergoing Valvular Heart Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2019-1051
Record Dates: First submitted 2019-12-12; First posted 2019-12-24 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Acute Kidney Injury
Keywords: Postoperative acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients are divided into 2 groups, who are administered IV Vitamin C or who are administered IV normal saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither participants, all care providers, investigators nor outcomes assessors know the treatment allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Participants in this group are administered IV normal saline.
  Interventions: Drug: Control (Normal saline)
- Vitamin C group (Experimental): Participants in this group are administered IV vitamin C diluted in normal saline.
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Vitamin C — Participants in "Vitamin C group" are administered IV vitamin C diluted in 100 cc normal saline 1 day before surgery, at rewarming during surgery, 3 hours after surgery, and every 6 hours thereafter until postoperative 24 hours.
  Arms: Vitamin C group
Drug: Control (Normal saline) — Participants in "Control group" are administered IV 100cc normal saline at the same timepoint as above.
  Arms: Control group

SUMMARY:
In cases of cardiac surgery or sepsis which cause inflammation, oxidative stress, endothelial injury and vasoplegia, serum vitamin C concentration is sharply decreased. The anti-inflammatory and anti-oxidant effects of vitamin C and the effects of reducing vasoconstrictor use have been demonstrated in patients with sepsis and septic shock, however, the foregoing effects have not been validated in patients undergoing cardiac surgery.

In this study, investigators investigate the effect of intravenous vitamin C on the incidence of acute renal injury after valvular heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years and undergoing elective valvular heart surgery whose preoperative acute renal failure score is ≥3 (moderate to severe risk).

Exclusion Criteria:

* Emergency operation
* Cardiogenic shock or ventricular-assist device (eg. ECMO, IABP)
* Severe chronic kidney disease (GFR(CKD-EPI) <30ml/min/1.73m2)
* Patients with past history of gout or renal stone or hyperoxaluria or cystinuria
* Hemolytic anemia due to pyruvate kinase deficiency or glucose-6-phosphate dehydrogenase deficiency
* Sicklemia or thalassemia
* Hemochromatosis
* Allergy to disodium ethylenediamine-tetraacetate or ascorbic acid
* Patients taking aspirin up to 3 days before surgery
* Patients taking antiepileptic drug or fluphenazine or steroid
* Patients taking vitamin C within a month of surgery
* Pregnant or lactating women
* Patients who cannot understand the informed consent (eg. Foreigner)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2020-03-24 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative acute kidney injury | Postoperative 7 days
  Compare the incidence of postoperative acute kidney injury between the Vitamin C group and the control group according to KDIGO guideline.

SECONDARY OUTCOMES:
Postoperative oxidative stress and vascular injury(Comparing the serum concentration) | Before anesthetic induction (Baseline)
  Compare the serum concentration of Malondialdehyde, Thrombomodulin before anesthetic induction and after CPB cessation.
Postoperative oxidative stress and vascular injury(Comparing the serum concentration) | 5 minute after CPB cessation
  Compare the serum concentration of Malondialdehyde, Thrombomodulin before anesthetic induction and after CPB cessation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine Anesthesia and Pain Research Institute, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No